CLINICAL TRIAL: NCT03749642
Title: Efficacy and Safety of Fixed-Dose Combination (FDC) Products Containing Trazodone and Gabapentin in Patients Affected by Painful Diabetic Neuropathy: Randomized, Controlled, Dose Finding Study.
Brief Title: Trazodone/Gabapentin Fixed Dose Combination Products in Painful Diabetic Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: Chiltern International Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 039(1)PO16357; 2018-000133-12 (EudraCT Number)
Record Dates: First submitted 2018-11-20; First posted 2018-11-21 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Painful Diabetic Neuropathy
Keywords: Trazodone; Gabapentin; Neuropathic pain; Placebo
MeSH Terms: conditions — Diabetic Neuropathies; Neuralgia | interventions — Trazodone; Gabapentin

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo and reference controlled, placebo unbalanced, double-dummy, dose finding, parallel group, multicentre, international, prospective study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The present study will be performed in double blind conditions. During the study neither the Investigator nor the patient will be aware of the treatment assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- trazodone/gabapentin 2.5/25 mg (Experimental): One capsule, three times a day, for 8 weeks. The total daily doses administered will be trazodone 7,5 mg and gabapentin 75 mg.
  Interventions: Drug: trazodone/gabapentin 2.5/25 mg
- trazodone/gabapentin 5/50 mg (Experimental): One capsule, three times a day, for 8 weeks.
  Interventions: Drug: trazodone/gabapentin 5/50 mg
- trazodone/gabapentin 10/100 mg (Experimental): One capsule, three times a day, for 8 weeks.
  Interventions: Drug: trazodone/gabapentin 10/100
- placebo (Placebo Comparator): Two capsules, three times a day, for 8 weeks.
  Interventions: Drug: Placebo oral capsule
- Gabapentin (Active Comparator): according to the following scheduling dosage regimen:
  * 100 mg (2 capsules) 3 times a day, from day 0 to day 6 (±1);
  * 300 mg (1 capsule) 3 times a day, from day 7 (±1) to day 13 (±1);
  * 400 mg (1 capsule) 3 times a day, from day 14 (±1) to day 20 (±1);
  * 300 mg (2 capsules) 3 times a day, from day 21 (±1) to day 55 (±2).
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: trazodone/gabapentin 2.5/25 mg — The total daily doses administered will be trazodone 7,5 mg and gabapentin 75 mg.
  Arms: trazodone/gabapentin 2.5/25 mg
Drug: trazodone/gabapentin 5/50 mg — The total daily doses administered will be trazodone 15 mg and gabapentin 150 mg.
  Arms: trazodone/gabapentin 5/50 mg
Drug: trazodone/gabapentin 10/100 — The total daily doses administered will be trazodone 30 mg and gabapentin 300 mg.
  Arms: trazodone/gabapentin 10/100 mg
Drug: Gabapentin — The total daily doses administered will be:
  * 600 mg from day 0 to day 6 (±1)
  * 900 mg from day 7 (±1) to day 13 (±1)
  * 1200 mg from day 14 (±1) to day 20 (±1)
  * 1800 mg from day 21 (±1) to day 56 (±2)
  Other Names: Neurontin
  Arms: Gabapentin
Drug: Placebo oral capsule — Two capsules, three times a day, for 8 weeks.
  Arms: placebo

SUMMARY:
The primary objective of the study is to collect preliminary information on the effect of three doses of trazodone/gabapentin FDC products on pain intensity in patients with painful diabetic neuropathy after 8-week treatment period.

DETAILED DESCRIPTION:
The present phase II study is designed to collect preliminary data on the efficacy and safety of trazodone/gabapentin Fixed-Dose Combination (FDC)products for treatment of patients affected by painful diabetic neuropathy in a randomized controlled clinical trial. Diabetic peripheral neuropathic pain represents an important therapeutic challenge as its pathophysiology is not yet fully understood and pain relief is still unsatisfactory. The pharmacological treatments, with exception to those targeted to the glycemic control, are symptomatic and their use is limited by not universal efficacy, side effects or by the development of tolerance. A wide variety of drugs, used both alone and in combination, has shown to significantly reduce neuropathic pain when compared with placebo in randomized controlled trials, even though pain relief remains inadequate for most of the patients.

In this contest, Angelini S.p.A is developing a fixed-dose combination medicinal product for the treatment of neuropathic pain containing low doses of active ingredients: trazodone, a widely used antidepressant drug, and gabapentin which is indicated for the treatment of neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patient of any ethnic origin between 18 and 75 years of age (limits included).
2. Neuropathic pain at feet/legs confirmed by Douleur Neuropatique 4 (DN4) score ≥ 4 at Screening Visit.
3. Patient with bilateral distal symmetrical polyneuropathy confirmed by Toronto Clinical Neuropathy Scoring System (TCNSS) score > 5 at Screening visit.
4. Pain persisting or taking pain medication for neuropathic pain for at least 3 months.
5. Diabetic patient (type 1 or 2 diabetes mellitus) with value of glycated haemoglobin ≤ 11% at Screening Visit and stable antidiabetic medication regimen for ≥30 days.
6. Patient who is currently not receiving treatment for diabetic neuropathic pain or patient who is receiving treatment, with drug/s other than gabapentin, and has completed the required washout.
7. Average daily pain score ≥ 4 based on the 11-point Numeric Rating Scale (NRS) at Visit 0, calculated from a minimum of four pain ratings in daily electronic device entries during the baseline period.
8. Women of childbearing potential must have a negative pregnancy test at Screening Visit and have to agree not to start a pregnancy from the signature of the informed consent up to thirty days after the last administration of the investigational product, using an appropriate birth control method, such as combined estrogen and progestogen containing hormonal contraception (e.g. oral, intravaginal, transdermal), progestogen-only hormonal contraception (e.g. oral, injectable, implantable), intrauterine device (IUD) or intrauterine hormone-releasing system (IUS) in combination with male condom, bilateral tubal occlusion, vasectomised partner, sexual abstinence.
9. Legally capable to give their consent to participate in the study (including personal data processing) and available to sign and date the written informed consent.

Exclusion Criteria:

1. Known hypersensitivity to trazodone or gabapentin or any excipients of the test drugs.
2. Any other form of non-diabetic distal symmetric polyneuropathy or any other pain condition that can impair the study endpoint (e.g. painful conditions where the intensity of pain is significantly more severe than the diabetic peripheral neuropathic pain).
3. Concomitant treatment with medications for pain management that could not be discontinued.
4. Concomitant treatment with potent CYP3A4 inhibitors (e.g. ketoconazole, ritonavir, indinavir) or drugs known to prolong QT interval.
5. Use of trazodone or gabapentin in the previous 3 months.
6. Known history of previous non-responder to gabapentin treatment.
7. Use of high dose morphine (e.g. > 120 mg/day) at the Screening Visit.
8. Clinically significant abnormalities on physical examination, vital signs, elettrocardiogram, laboratory tests at Screening Visit that in the opinion of Investigator would compromise patient's participation in the study.
9. Active foot ulcer or previous major limb amputation.
10. Concurrent heart failure ≥ 4 class according to New York Heart Association (NYHA) or myocardial infarction or angioplasty or by-pass graft procedures within the past 6 months.
11. Patient with increased risk of Torsade de Pointes (e.g. family history of long QT syndrome) or QTcF value higher than 450 msec (male) and QTcF value higher than 470 msec (female) at Screening Visit.
12. Transient ischemic attack or cerebral vascular accident within the past 6 months.
13. Glomerular Filtration Rate value < 50 ml/min calculated with Modification of Diet in Renal Disease formula.
14. Significant liver disease, defined as known active hepatitis or elevated liver enzymes over 3-fold the upper normal limit of laboratory normal ranges.
15. Patient with latent or known hereditary problems of galactose intolerance or the Lapp lactase deficiency or glucose-galactose malabsorption.
16. Positive urine drug screen for Central Nervous System active drugs (cocaine, opioids, amphetamines and cannabinoids) at Screening Visit.
17. Positive present history of glaucoma.
18. Hyperthyroidism, even if pharmacologically corrected.
19. Significant mental disorders.
20. Suicide risk score ≥ 2 on question 9 of the Beck Depression Inventory-II (BDI-II) at Screening visit or Visit 0.
21. History of epilepsy or seizure events other than a single childhood febrile seizure.
22. History of alcohol or psychoactive substance abuse or addiction.
23. Use of neurological device (e.g. neurostimulation devices, etc).
24. Women during pregnancy or lactation period.
25. Inability to comply with the protocol requirements, instructions or study-related restrictions (e.g. uncooperative attitude, inability to return for study visits, improbability of completing the clinical study, etc).
26. Subject involved in the conduct of the study (e.g. Investigator or his/her deputy, first grade relatives, pharmacist, assistant or other personnel, etc).
27. Participation to an interventional clinical trial within 3 months prior to Screening Visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2018-11-22 (Actual); Primary Completion 2020-06-06 (Actual); Study Completion 2020-06-06 (Actual)

PRIMARY OUTCOMES:
Change of the average daily pain score based on the 11-point Numeric Rating Scale (NRS). | Baseline - Day 56
  The NRS is based on a 11-point from 0 for [no pain] to 10 [worst possible pain].

SECONDARY OUTCOMES:
Change of the average daily pain score based on the 11-point Numeric Rating Scale (NRS). | Baseline - Days 7, 14, 21, 28, 42
  The NRS is based on a 11-point from 0 for [no pain] to 10 [worst possible pain].
Percentage of responder patients | Baseline - Day 56
  Responder patients are defined as ≥30% and ≥50% reduction from baseline of the average daily pain score based on the 11-point NRS.
Change of the average daily pain score based on the 11-point NRS between gabapentin and placebo as assay sensitivity. | Baseline - Day 56
  The NRS is based on a 11-point from 0 for [no pain] to 10 [worst possible pain].
Change of Brief Pain Inventory Short Form (BPI-SF) items 3, 4, 5, 6, 8 and 9 score. | Baseline - Days 28, 56
  The BPI-SF is a numeric rating scale that assesses the severity of pain, its impact on daily functioning and other aspects of pain (e.g. location of pain, relief from medications). Items use a 0-10 numeric rating scale anchored at zero for "no pain" and 10 for "pain as bad as you can imagine" for Severity, and "does not interfere" to "completely interferes" for Interference.
Change of Neuropathic Pain Symptom Inventory (NPSI) total score. | Baseline - Days 28, 56
  The NPSI is a self-questionnaire specifically designed to evaluate the different symptoms of neuropathic pain: It includes 10 descriptors plus two temporal items that allow discrimination and quantification of five distinct clinically relevant dimensions of neuropathic pain syndromes.
Change of Beck Depression Inventory - Second Edition (BDI-II) | Baseline - Days 28, 56
  The BDI-II consists of 21 items to assess the intensity of depression in clinical and normal patients. Each item is a list of four statements arranged in increasing severity about a particular symptom of depression and scored from 0 to 3.
Change of Hospital Anxiety and Depression Scale (HADS). | Baseline - Days 28, 56
  The HADS is used to assess the level of anxiety and depression that a patient is experiencing. This is 14-item scale: seven related to the anxiety and seven to depression. Each item is scored from 0 to 3.
Change of Insomnia Severity Index (ISI). | Baseline - Days 28, 56
  The ISI is a 7-item self-reported instrument measuring the patient's perception of his/her insomnia.Total score ranges from 0-28 and the following categorization is applicable: 0-7 = absence of insomnia; 8-14 = subthreshold insomnia; 15-21 = moderate insomnia; 22-28 = severe insomnia.
Change of Euroqol-5D-5L (EQ-5D-5L) | Baseline - Days 28, 56
  The EQ-5D-5L consists of the EQ-5D descriptive system (five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression assessed as no problems, slight problems, moderate problems, severe problems and extreme problems) and the EQ visual analogue scale (where the patient self-rates his/her health on a vertical visual analogue scale from 'The best health you can imagine' to 'The worst health you can imagine').
Clinical Global Improvement or Change (CGI-C). | Baseline - Days 28, 56
  CGI-C provides a global rating of patient's Improvement and scores range from "0 - not assessed" through to "7 - very much worse".
Frequency of adverse events | 65 days
  Monitoring of the treatment related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Solomon Tesfaye, MD, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (30):
- Czechia (7):
  - Neurosanatio s.r.o., Litomyšl, 570 01
  - Cerebrovaskulární poradna, s.r.o., Ostrava - Poruba, 70800
  - Nemocnice Pardubického kraje a.s. Pardubická nemocnice Neurologická klinika, Pardubice, 532 03
  - Diabetologická ambulance Milan Kvapil s.r.o., Praha 4, 149 00
  - Axon Clinical s.r.o, Praha 5, 15000
  - FORBELI s.r.o., Praha 6, 160 00
  - Clintrial s.r.o., Praha, 100 00
- France (4):
  - Fondation Hôtel Dieu Groupe SOS Service de Diabétologie, Le Creusot
  - GHR MSA - Hôpital Emile Muller Service de Diabétologie-Endocrinologie-Nutrition, Mulhouse
  - CHU de Nantes - Hôpital Guillaume-et-René-Laënnec Clinique d'Endocrinologie, maladies métaboliques et nutrition CIC Endocrino - Nutrition - UF 7015, Nantes Cedex 144 093
  - Centre de Recherche Clinique G.H.M les Portes du Sud Departement d'Endocrinologie, Vénissieux
- Poland (13):
  - Centrum Badań Klinicznych PI-House, Gdansk, 80-546
  - Silmedic Sp. z o.o., Katowice, 40-282
  - Pro Familia Altera Poradnia Wielospecjalistyczna, Katowice, 40-648
  - Medyczne Centrum Diabetologiczno-Endokrynologiczno-Metaboliczne DIAB-ENDO-MET, Kraków, 31-261
  - NZOZ Neuromed M. i M. Nastaj Sp. P., Lublin, 20-064
  - Instytut Medycyny Wsi im. Witolda Chodźki Klinika Diabetologii, Lublin, 20-090
  - Centrum Medyczne HCP Sp. z o.o., Poznań, 61-485
  - RCMed Oddział Sochaczew, Sochaczew, 96-500
  - Nasz Lekarz Przychodnie Medyczne, Toruń, 87-100
  - Medycyna Kliniczna, Warszawa, 00-874
  - Instytut Diabetologii, Warszawa, 04-736
  - WroMedica I. Bielicka, A. Strzałkowska s.c., Wrocław, 51- 685
  - Centrum Badań Klinicznych Ośrodek Badań Wczesnej Fazy, Wrocław, 51-162
- United Kingdom (6):
  - Medical Innovation Development and Research Unit (MIDRU) Heartlands Hospital, Birmingham
  - Diabetes Centre Wythenshawe Hospital, Manchester
  - Manchester Clinical Research Facility Manchester Royal Infirmary, Manchester
  - Diabetes Centre George Eliot Hospital NHS Trust, Nuneaton
  - Lancashire Clinical Research Facility The Avondale Unit Royal Preston Hospital, Preston
  - Clinical Research Facility Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tesfaye S, Saravanan P, Ehler E, Zinek K, Palka-Kisielowska I, Nastaj M, Serusclat P, Lipone P, Vergallo A, Quarchioni E, Calisti F, Comandini A, Cattaneo A. Efficacy and Safety of Trazodone and Gabapentin Fixed-Dose Combination in Patients Affected by Painful Diabetic Neuropathy: Randomized, Controlled, Dose-Finding Study. Pain Ther. 2024 Aug;13(4):987-1006. doi: 10.1007/s40122-024-00624-3. Epub 2024 Jun 24. PMID 38914876